CLINICAL TRIAL: NCT04605016
Title: Clinical Performance of Dental Implants With Hydrophilic or Hydrophobic Surfaces in Single Posterior Edentulous Spaces: a Randomized Clinical Trial
Brief Title: Clinical Performance of Dentals Implants With Hydrophilic or Hydrophobic Surfaces
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidade Federal de Goias (Other)
Responsible Party: Principal Investigator, Cláudio Rodrigues Leles, Full Professor, Universidade Federal de Goias
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PI04791-2020
Record Dates: First submitted 2020-10-15; First posted 2020-10-27 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Tooth Loss
Keywords: single tooth gap; missing tooth
MeSH Terms: conditions — Tooth Loss; Anodontia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydrophilic surface implants (Experimental)
  Interventions: Device: Hydrophilic surface implants
- Hydrophobic surface implants (Active Comparator)
  Interventions: Device: Hydrophobic surface implants

INTERVENTIONS:
Device: Hydrophilic surface implants — A dental implant with hydrophilic surface will be placed and restored in single-tooh gaps of the posterior region of the mandible or maxilla.
  Other Names: Neodent Helix Grand Morse® Acqua
  Arms: Hydrophilic surface implants
Device: Hydrophobic surface implants — A dental implant with hydrophobic surface will be placed and restored in single-tooh gaps of the posterior region of the mandible or maxilla.
  Other Names: Neodent Helix Grand Morse® Neoporos
  Arms: Hydrophobic surface implants

SUMMARY:
The aim of the study is to compare longitudinally the clinical performance of dental implants with different surfaces placed in single tooth gaps at the posterior maxilla and mandible of adults. It is a randomized clinical trial, in which participants will be randomly allocated to two groups: test group (implants with hydrophilic surface) and control group (implants with hydrophobic surface). The null hypothesis is that the implant stability quotient of hydrophilic and hydrophobic dental implants show a similar progression after placement in posterior tooth gaps.

ELIGIBILITY:
Inclusion Criteria:

* Present single or multiple intercalated untreated tooth gaps in the posterior region of the mandible or maxilla;
* Agree to participate in the study by signing the informed consent form.

Exclusion Criteria:

* Unavailability for participation or signs that they could not comply with the schedule of follow-up visits;
* Presence of general and/or local contraindications that could prevent the surgical procedure for implant placement;
* Presence of conditions that may interfere with the prognosis, such as current treatment with bisphosphonates or report of use for less than 2 years, presence of rheumatic diseases, among others;
* Absence of the minimum bone quantity of 8 mm in length and 3.75 mm in diameter for installation of an implant in the tooth gap;
* Absence of a mesio-distal space of at least 4.6 mm in the single tooth gap required to place the surgical guide;
* Do not present a mouth opening of at least 12mm required for the proper of the guided surgical kit together with the surgical guide;
* Do not present a band of keratinized tissue favorable for maintaining peri-implant health.
* Present motor difficulties that compromise adequate oral hygiene.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-09-11 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Change of implant stability | 10 time-points will be considered and divided in two phases: surgical and prosthetic. The last measure will occur 1 year after the placement of the definitive implant restoration.
  Implant stability was set as the primary outcome. The implant stability quotient (ISQ) will be measured using a portable device called Osstell ISQ (Osstell Mentor, Integration Diagnostics, Göteborg, Sweden).

SECONDARY OUTCOMES:
Implant success | Assessed at the 12-month follow-up visit.
  Each implant will be assessed according to the health scale of the International Congress of Oral Implantologists (ICOI-Pisa health scale). After clinical assessment, each implant will be classified as 'success', 'satisfactory survival', 'compromised survival' or 'failure'.
Periimplant bone level | Radiographs will be obtained at 4 time points: immediately after implant placement, at the session of the provisional prosthesis installation, and at the 6 and 12-month follow-up visits after the delivery of the definitive prosthesis.
  Periapical radiographs will be obtained and the periimplant bone level will be measured and compared longitudinally.
Condition of the periimplant soft tissues | 15-days, 6- and 12-month follow-up visits after delivery of the definitive prosthesis.
  The following parameters will be assessed clinically: presence/absence of bleeding on probing, probing depth, and presence/absence suppuration.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry of the Federal University of Goias, Goiânia, Goiás, Brazil